

March 23, 2023 

### Informed Consent/Authorization for Participation in Research

TITLE: A Phase II Study to evaluate the efficacy

and safety of pembrolizumab in

combination with mitotane in patients with

advanced adrenocortical carcinoma

PROTOCOL NO.: 2022-0705

SPONSOR: Merck Sharp & Dohme

**INVESTIGATOR:** Mouhammed A. Habra, MD

STUDY-RELATED

PHONE NUMBER(S): 713-792-2841

713-792-2121 (24 hours)

Participant's Name

Medical Record Number

# **Key Information**

The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

## Why am I being invited to take part in a research study?

You are invited to take part in a research study because you have adrenocortical carcinoma (ACC).

## What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.




## Why is this research being done?

ACC is a rare cancer with limited treatment options. Mitotane is the only FDA-approved drug that is considered standard of care for this disease. Immunotherapy has recently been studied as a way of enhancing the effects of mitotane. Pembrolizumab is a form of immunotherapy that has been studied in adrenal cancer patients, but it is not FDA-approved for the treatment of the disease. Its use in this study is investigational.

The goal of this clinical research study is to learn if adding pembrolizumab to mitotane can help to control ACC. The safety of this drug combination will also be studied.

## How long will the research last and what will I need to do?

You are expected to be in this research study for up to 2 years.

You will be asked to receive infusions of pembrolizumab and take mitotane by mouth during the study. You will also have study visits at which various tests and procedures will be performed, such as blood draws and imaging scans. You will also have optional tumor biopsies, if you agree to them. They are not required.

If you the study doctor thinks it is in your best interest, you may be able to continue receiving mitotane after 2 years. They will discuss this with you.

More detailed information about the study procedures can be found under "What happens if I agree to be in this research?"

## Is there any way being in this study could be bad for me?

Mitotane is known to cause adrenal insufficiency (low adrenal hormone level) in most patients that receive it. This often requires steroid replacement. Mitotane can also cause diarrhea, upset stomach, abnormal liver function, and fatigue.

Pembrolizumab is usually well tolerated, but because it enhances the immune system's response to cancer, it can cause side effects that vary depending on the involved organs. For example, if the immune system is enhanced to attack the bowels, then patients may have diarrhea, bloody stools, and abdominal discomfort. While many of these side effects are manageable, occasional and unpredictable life-threatening effects can occur.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"




## Will being in this study help me in any way?

It cannot be promised that there will be any benefits to you or others from your taking part in this research. However, the study drugs may help to control the disease. Future patients may benefit from what is learned.

### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

Instead of being in this research study, your choices may include other available treatments for cancer, such as chemotherapy or targeted therapy. You may be eligible for other cancer research studies. You may receive treatment for pain or other symptoms only. These alternative treatments have risks and benefits that may be the same or different than those in this research study. The study doctor can discuss these alternative treatments, including their risks and benefits with you.


## **Detailed Information**

The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to if I have questions or concerns?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at 713-792-2841. You may talk to them at (713) 792-6477 or IRB\_Help@mdanderson.org if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

#### How many people will be in this study?

It is expected about 50 people at MD Anderson will be enrolled in this research study.

#### What happens if I agree to be in this research?

#### **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible:

- You will have a physical exam.
- Blood (about 2-3 tablespoons) will be drawn for routine tests. If you are already receiving mitotane, your mitotane levels will be checked.
- You will have an EKG to check your heart function.
- You will have imaging scans (CT, MRI, and/or PET scans) to check the status of the disease.
- If you can become pregnant, your blood or a urine sample will be used for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

#### **Study Drug Administration**

If you are found to be eligible to take part in this study, you will first have a Lead-in phase in which you receive only mitotane. This will be 4 weeks long in most participants. You will then begin receiving pembrolizumab. If you have already been




receiving mitotane for at least 4 weeks when you begin the study, you do not have to have the Lead-in phase.

You will take mitotane by mouth every day at about the same time. It should be taken with food. If it is missed by more than 6 hours or vomited, do not replace the dose. Wait until your next dose.

You will receive pembrolizumab by vein every 6 weeks, over about 30 minutes each time.

#### **Study Visits**

During the Lead-in phase, you will have standard tests and procedures to check your health. This will be discussed with you. After that, each study cycle will be 6 weeks (42 days) long.

#### On Day 1 of each cycle:

- You will have a physical exam.
- Blood (about 2-3 tablespoons) will be drawn for routine tests and to check your mitotane levels.
- You will have imaging scans to check the status of the disease (every evennumbered cycle only [Cycles 2, 4, 6, and so on]).
- If you can become pregnant, your blood or a urine sample will be used for a pregnancy test.

#### **End-of-Dosing**

After you stop receiving the study drugs:

- You will have a physical exam.
- Blood (about 2-3 tablespoons) will be drawn for routine tests and to check your mitotane levels.

### Follow-Up

You will be called every 3 months and asked about how you are doing. Each call should take on average 5-10 minutes.

If you left the study for reasons other than the disease getting worse, you will continue to have imaging scans every 12 weeks to check the status of the disease.

# What are my responsibilities if I take part in this research?

You will need to tell and get approval from the study team if you would like to participate in other ongoing research that does not conflict with the study intervention and procedures. While on this study, it is not allowed to receive other anti-cancer treatment or enroll in other clinical studies that treat cancer. You will need to tell the study team to end your participation in this study before enrolling in other clinical trials or receiving other cancer treatments.




If you take part in this research, you will be responsible for telling the study team about any symptoms or side effects you have, following study directions, and coming to all study appointments (or contacting the study team to reschedule).

## What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you.

If you decide to leave the research, there is possibility of tumor growth in case the treatment is effective and stopped. If you decide to leave the research, contact the study doctor so that the study doctor can process the end of your study participation and the needed tests and procedures if needed to ensure a smooth end of the study participation. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

# Is there any way being in this study could be bad for me? (Detailed Risks)

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

#### **Mitotane Side Effects**

# Common (occurring in more than 20% of patients)

| • | depression | • | loss of appetite | • | nausea |
|---|------------|---|------------------|---|----------|
| • | dizziness | • | diarrhea | • | vomiting |

## Occasional (occurring in 3-20% of patients)


#### skin rash

#### Frequency unknown

- flushing
- high blood pressure
- low blood pressure (possible dizziness/fainting)
- fever
- difficulty walking
- fatigue
- confusion
- difficulty forming or speaking words
- mental status change
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)

- high blood levels of fat (possible heart disease and/or stroke)
- changes in hormone levels (including low levels of testosterone)
- enlarged breasts in males
- blood in the urine
- bladder inflammation with bleeding (possible pain and/or urge to urinate)
- ovarian cysts (fluid-filled lumps)

- low white blood cell count
- increased risk of bleeding
- liver damage
- abnormal liver tests (possible liver damage)
- pain
- weakness
- blurry vision
- cataracts (clouding of the lens of the eye)
- double vision
- eye damage causing vision problems
- damage to the retina (possible vision loss)
- abnormal kidney test (possible kidney damage)

There are currently no known side effects occurring in **fewer than 3% of patients**.

## **Pembrolizumab Side Effects**

Common (occurring in more than 20% of patients)




- fatigue
- fever
- skin rash and/or itching
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- high blood sugar (possible diabetes)
- high blood levels of fat (possible heart disease and/or stroke)
- loss of appetite
- nausea
- constipation
- diarrhea
- abdominal pain

- low blood cell counts (red, white, platelets)
- abnormal liver test (possible liver damage)
- pain
- abnormal kidney test (possible kidney damage)
- cough
- difficulty breathing

Pembrolizumab may commonly cause low blood cell counts (red, white, and/or platelets):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life- threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.

#### Occasional (occurring in 3-20% of patients)

- swelling (face/arm/leg)
- inflammation of the tissue around the heart (possible chest pain)
- irregular heartbeat
- headache
- confusion
- patches of skin color loss
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- overactive thyroid gland (possible weight loss, diarrhea, mood swings, difficulty sleeping, heart rate changes, and/or sweating)
- low blood sugar
- weight loss
- fluid in the abdomen
- blood in the urine
- vomiting
- abnormal liver test (possible yellowing of the skin and/or eyes)

- weakness
- nerve damage (possible numbness, pain, and/or loss of motor function)
- difficulty breathing (possibly due to lung inflammation)
- flu-like symptoms
- infusion reaction (possible dizziness, low blood pressure, nausea, pain, and/or difficulty breathing)

#### **Frequency Unknown**

heart failure
abnormal connections
blockage in the lung




- heart attack
- build-up of fluid around the heart (possible heart failure)
- or passageways between organs or vessels
- bleeding in the rectum and/or uterus

(possible pain and/or shortness of breath)

- nosebleed
- coughing up blood

#### Rare but serious (occurring in fewer than 3% of patients)

- low blood pressure (possible dizziness/fainting)
- heart inflammation
- build-up of fluid in the tissue around the heart
- blood vessel inflammation (possible bleeding, skin rash, numbness/weakness, fever, weight loss, fatigue, and/or bruising, depending on where the inflammation occurs)
- seizure
- immune system damage to the nervous system (causing muscle weakness, numbness and/or paralysis)
- spinal cord inflammation (possible pain, weakness, loss of feeling or movement, and/or paralysis)
- brain inflammation (possible paralysis and/or coma)
- shedding, scaling and/or inflammation of the skin (possible fatal loss of bodily fluids)
- large skin blisters
- very severe blistering skin disease (loss of

- low hormone blood levels (possible weakness, bone changes, and/or cramping)
- hormonal deficiency that affects the body's ability to control blood pressure and react to stress
- pituitary gland inflammation (possible headaches)
- inflammation of the thyroid gland (possible tenderness in the neck)
- diabetes requiring insulin
- severe high blood sugar due to uncontrolled diabetes
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)
- inflammation of the pancreas (possible abdominal pain)
- anemia due to destruction of red blood cells
- liver damage (hepatitis)
- inflammation/scarring of the bile ducts (tubes that carry digestive fluid that is made in the

- inflammation inside the eye (possible vision problems)
- kidney inflammation (possible kidney damage/failure)
- kidney failure
- build-up of fluid around the lungs
- immune response that causes the body to attack itself (possible organ damage)
- multi-organ disease causing lesions, most often in the lungs (sarcoidosis)
- immune response (causing muscle weakness)
- immune system reaction (possible fever, jaundice, liver/spleen enlargement, irritability, and/or seizures)
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- Vogt Koyanagi Harada syndrome -- pigmented tissue (possible eye pain/swelling and changes in vision, hearing loss, and/or white patches on the




| large portion of skin | liver), which may cause | skin) |
|---------------------------|-------------------------|-------|
| and/or with ulcers of the | liver damage, stomach | |
| skin and digestive tract) | pain, yellowing of the | |
| | skin/eyes, fatigue, | |
| | and/or itching | |

If you have a solid tumor type and you have an organ transplant, pembrolizumab may increase your risk for the transplant to be rejected by your body.

Pembrolizumab works by boosting the immune system. This may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue. These side effects can affect more than one of your normal organs and tissues at the same time.

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.




CT scans send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

A **PET scan** may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort, or the scanning will be stopped.

The PET scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**.

In addition to these risks, this research may hurt you in ways that are unknown. These may be a minor inconvenience or may be so severe as to cause death.

You will be told about any new information that may affect your health, welfare, or choice to stay in the research.

#### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Females: You must use highly effective birth control, such as a progesterone only implant, an intrauterine hormone-releasing system (IUS), an intrauterine device (IUD), or bilateral tubal ligation ("tubes tied"). A vasectomized partner is a highly effective birth control method if this partner is your only male sexual partner and the absence of sperm has been confirmed. If not, an additional highly effective method of birth control should be used.




If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

Males: You should use condoms while on study, and any female partners should also use one of the methods of birth control described for females above.

Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

# Will it cost anything to be in this study? Will I be paid to be in this study?

Pembrolizumab will be provided at no cost to you on this study, but you and/or your insurance provider will be responsible for the cost of pembrolizumab administration. You and/or your insurance provider will be responsible for the costs of mitotane.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

You will not receive any compensation for taking part in this study.

# What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who need to review this information. Complete secrecy cannot be promised. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

Any personal information that could identify you will be removed or changed before data are shared with other researchers or results are made public.

The sponsor, monitors, auditors, the IRB, and the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.




Federal law provides additional protections of your medical records and related health information. These are described below.

### Will my data or samples be used for future research?

Your personal information and/or samples are being collected as part of this study. These data may be used by researchers at MD Anderson and Merck, or shared with other researchers and/or institutions for use in future research. Samples may be used by researchers at MD Anderson.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the MD Anderson IRB before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

If identifiers are removed from your identifiable private information or identifiable samples that are collected during this research, that information or those samples could be used for future research studies or shared with another researcher for future research studies without your additional informed consent.

## Can I be removed from the research study without my permission?

The person in charge of the research study or the sponsor can remove you from the research study without your approval. Possible reasons for removal include side effects of therapy, concerns about compliance with study procedures and requirements, or worsening of disease, among others.

# What happens if I get hurt from being in this study?

If you get sick or hurt and it is related to your participation in this study, you will be given care at MD Anderson (if you are at the clinic when you are sick or hurt). If you get hurt or sick and you are not at the clinic (for example, you are at home or at another doctor's office):

- call your personal doctor right away (or in an emergency, call 911)
- tell your personal doctor or ER staff that you are in this study (try to give them a copy of this consent form or show them your participant card)
- call the study doctor (Dr. Habra, at 713-792-2841) or the 24-hour phone number (713-792-2121)

You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. Costs of treatment received because you were hurt or sick will be billed to you or your insurance company. No other form of payment is available.




In case of you were hurt or got sick during the study including potential side effects of treatments, you or/and your insurance carrier will pay for the treatment you received . A financial counselor will be made available to you after the injury or illness is reported.

You may also contact the MD Anderson IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

#### What else do I need to know?

This research is being funded by Merck Sharp & Dohme.

MD Anderson may benefit from your participation and/or what is learned in this study.

Your information and samples (both identifiable and de-identified) may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

Most tests done on samples in research studies are only for research and have no clear meaning for health care. If the research with your identifiable information or samples gives results that do have meaning for your health, the researchers will not contact you to let you know what they have found. If the researchers return genetic test results to you, it may be because they think you could have a health risk and want to recommend that the test should be re-done by a certified clinical laboratory to check the results. If this happens, then you may want to get a second test from a certified clinical laboratory, consult your own doctor, or get professional genetic counseling. You may have to pay for those additional services yourself.

This research study involves genetic testing. The Genetic Information Nondiscrimination Act (GINA) prohibits health insurers or health plan administrators from requesting or requiring genetic information of you or your family members, or using such information for decisions regarding your eligibility for insurance or your premiums. However, this law does <u>not</u> provide the same protection for disability, life insurance, or long-term care insurance. GINA also prohibits most employers (with 15 employees or more) from using genetic information when making decisions on your employment, including decisions related to hiring, firing, promotion, pay, and job assignments. Please contact the study doctor if you would like more information about GINA and how it protects you from genetic discrimination.

Genetic research may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment.




## **Optional Procedures for the Study**

You do not have to agree to the optional procedure in order to take part in this study. There are no benefits to you for taking part in the optional procedure. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedure.

**Optional Procedure #1:** If you agree, you will have up to 3 optional tumor biopsies if the study doctor thinks they are accessible. These will be performed at screening, on Day 1 of Cycle 4, and then if at any time the disease gets worse.

**Optional Procedure Risks:** Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES Circle your choice of "yes" or "no" for each of the following optional procedures:

Optional Procedure #1: Do you agree to have tumor biopsies?

YES NO

# Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Merck Sharp & Dohme, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study, and/or licensees of the study technology
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.




The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI, and it may be re-disclosed.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.




#### **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| PRINTED NAME OF PARTICIPANT | |
| LEGALLY AUTHORIZED REPRESENTATIVE (LAR) | |
| The following signature line should only be filled out when the partic the capacity to legally consent to take part in the study and/or sign the or her own behalf. | |
| SIGNATURE OF LAR | DATE |
| PRINTED NAME and RELATIONSHIP TO PARTICIPANT | |
| WITNESS TO CONSENT | |
| I was present during the explanation of the research to be performed protocol. | I under this |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT | |
| I have discussed this research study with the participant and/or his o | |
| representative, using language that is understandable and appropria have fully informed this participant of the nature of this study and its and risks and that the participant understood this explanation. | |
| PERSON OBTAINING CONSENT | DATE |


# PRINTED NAME OF PERSON OBTAINING CONSENT




## **TRANSLATOR**

| I have translated the above | informed consent as written (without add | ditions or |
|---|---|---|
| subtractions) into | and assisted | and assisted the people |
| (Nam | e of Language) | guage) |
| obtaining and providing conscious consent process for this part | sent by translating all questions and resplicipant. | oonses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| | translator was a member of the researc<br>an the translator, must sign the witness | ` |